CLINICAL TRIAL: NCT05367479
Title: The Effect of Peri-operative Antibiotic Class on Microbiome Changes After Roux-en-Y Gastric Bypass
Brief Title: Antibiotics, Gastric Bypass, and the Microbiome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Tammy Kindel, MD, PhD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO00030985
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Obesity, Morbid; Hypertension; Bariatric Surgery Candidate
Keywords: gut microbiome
MeSH Terms: conditions — Obesity, Morbid; Hypertension | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cefazolin (Active Comparator): standard of care as a pre-operative antibiotic given with 60 minutes of incision before gastric bypass surgery. given intravenous as a single dose, weight based.
  Interventions: Drug: Antibiotic
- Clindamycin (Active Comparator): also standard of care alternative as a pre-operative antibiotic given with 60 minutes of incision before gastric bypass surgery. given intravenous as a single dose, weight based.
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — Peri-operative, intravenous antibiotic for surgical site infection

SUMMARY:
This study randomizes patients to two commonly used peri-procedural antibiotics after gastric bypass with the pre and post-operative collection of stool samples, to identify significant differences in relative abundances of gut microbiota phyla, genera and species between the two antibiotic groups used. Gastric bypass may beneficially affect hypertension by altering the post-operative microbiome and specific antibiotics can further enhance the resolution rate by improving microbial diversity and richness.

DETAILED DESCRIPTION:
Eligible patients will be reviewed to meet inclusion criteria. Patients will be approached for enrollment at their pre-operative clinic appointment. If patients agree, consent will be signed.

Demographics will be collected on all patients including past medical, surgical and obesity history. Blood pressure will be recorded in the office, hypertensive medication record reviewed, post-operative follow-up and stool samples will be collected at 5 visits (V1-V5): 2 weeks pre-op, day of surgery, 2 weeks post-op, and 3 months post-op. Patients will be randomized at the time of surgery to receive intravenous cefazolin or clindamycin (weight-based dosing) as a pre-operative antibiotic within 60 minutes of incision time. Both antibiotics are routinely used as a single intravenous pre-operative dose for surgical site infection prophylaxis during Roux-en-Y gastric bypass and does not alter the standard of care. In routine care, clindamycin is given when there is a cefazolin allergy. Vancomycin is given if there is an allergy to both. We have a protocol that all bariatric surgeons follow rather than preference. There should be equipoise regarding the risk of a skin, superficial or deep surgical site infection between the two choices.

Hypertension will be considered resolved when the blood pressure is <140/90 without medication. Data points for collection were chosen to identify both short and long-term changes in the microbiome as well as assess for changes in the microbiome related to dietary modifications required with surgery.

Stool samples will be collected from participants in this study. Stool samples will be collected at the convenience of the participant at time points designated in the study design. The participant will be given a stool sample kit(s) to take home during the time of consent. The stool sample will be received by the research laboratory at a follow-up visit, or returned via FedEx with materials supplied in the stool collection kit. Following receipt in the laboratory, the stool samples will be stored in Dr. Kindel's lab (4th floor CRI) at -80 degrees where they will later undergo bacterial genomic DNA and RNA isolation using standardized techniques and later analysis for 16S and metagenomic sequencing analysis.

ELIGIBILITY:
Inclusion Criteria: Patients who are approved for a primary RYGB at MCW's bariatric surgery program as treatment for morbid obesity and obesity-associated co-morbidities. Patients will be eligible who are: 1.) female or male 2.) 18-70 years of age, 3.) hypertensive

Exclusion Criteria: Patients are ineligible if they: 1.) have a diagnosis of cirrhosis, 2.) are taking antibiotics, probiotics, or immune modulating medications for one month prior to or after surgery, 3.) have a history of bowel resections, inflammatory bowel disease and/or celiac disease, 4.) have a life-threatening reaction to penicillin/cephalosporins or clindamycin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
operational taxonomic units | 3 months postoperatively
  a distinct bacterial community

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No